CLINICAL TRIAL: NCT01393405
Title: Randomized, Double Blind, Prospective Trial Investigating the Efficacy of Methotrexate in Induction and Maintenance of Steroid Free Remission in Ulcerative Colitis (MEthotrexate Response In Treatment of UC - MERIT-UC)
Brief Title: Methotrexate in Induction and Maintenance of Steroid Free Remission in Ulcerative Colitis
Acronym: Merit-UC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hans Herfarth, MD, PhD, Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-2044; 1U01DK092239-01 (NIH)
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate (Active Comparator): 25 mg MTX sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Placebo sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Induction period (week 1-16) (Open label):
  25 mg MTX sq once weekly + Steroid taper + 1 mg folic acid daily
  Maintenance period (week 17-48) (Randomization):
  25 mg MTX sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine or Placebo sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine
  Other Names: Placebo

SUMMARY:
There are fewer therapeutic options for patients with active ulcerative colitis (UC) compared to patients with active Crohn's disease (CD) and the investigators are facing a persistent unmet need for additional effective and affordable therapies for patients with UC. Methotrexate (MTX) 25 mg once weekly administered subcutaneously (sq) or intramuscularly (im) is an efficient therapy to induce and maintain steroid free remission in patients with CD. To evaluate the efficacy of a similar approach in patients with active ulcerative colitis the investigators conduct a double-blind, placebo controlled, randomized, multicenter, parallel group trial to investigate the safety and efficacy of 25 mg MTX applied subcutaneously once weekly in patients with active UC, who either failed 5-ASA therapy, or are steroid dependent or are intolerant or not responding to azathioprine/6-mercaptopurine therapy or have no response/ lost response to infliximab prior to the study inclusion. The study is designed as a drug withdrawal trial and includes two periods, the Induction Period (week 0-16) and the Maintenance Period (week 17-48). In the open label Induction Period every patient will receive a steroid taper, MTX 25 mg sq once weekly + daily folic acid 1 mg tablets for the induction of clinical response or remission. Patients responding to the open label MTX therapy and being off steroids between week 12-16 will be randomized at week 16 1:1 to Placebo sq once weekly + daily folic acid 1 mg tablets + 2.4 g mesalamine or to MTX 25 mg sq once weekly + daily folic acid 1 mg tablets+ 2.4 g mesalamine. The Specific Aims of the trial are: i) To evaluate the safety and tolerability of 25 mg MTX applied sq once weekly over a time period of 48 weeks; ii) To evaluate the relapse-free survival of MTX maintenance therapy compared to placebo over a time period of 32 weeks; iii) To evaluate the efficacy of MTX over a time period of 16 weeks to induce steroid free remission; iiii) To establish a DNA, plasma and serum library to enable the evaluation of clinical and pharmacogenomic models to predict the response to MTX therapy in patients with UC. With 25-30 participating centers actively enrolling, the investigators anticipate to complete enrollment for this study in a time period of 3 years. Completion of this trial will define the therapeutic value of MTX in UC, potentially changing the current therapeutic strategy in UC.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Man or woman between 18 and 70 years of age.
* UC diagnosed by routine clinical, radiographic, endoscopic, and pathological criteria.
* Active UC with a Mayo score of 6 to 12 points and moderate-to severe active disease on sigmoidoscopy (Mayo endoscopic subscore of at least 2)

and at least ONE of the following criteria:

* Steroid dependent UC *
* Primary failure or loss of response to an anti-TNF (infliximab, adalimumab, golimumab) in the past
* Primary failure or loss of response to vedolizumab in the past
* Intolerance/failure of azathioprine/6-MP therapy in the past
* Failure of 5-ASA therapy

  * Steroid dependence is defined as a clinical response to treatment with prednisone 40 to 60 mg/day and relapse within 30 days after prednisone treatment was completed or as a requirement for a daily dosage of not less than 10 mg of prednisone and impossibility of weaning the patient off steroid without clinical relapses (two attempts to discontinue the medication within the preceding six months of the start of the study).

Exclusion Criteria:

* Failure to respond to 40 mg of prednisone or higher/day in the last 2 weeks before inclusion
* Concomitant use of azathioprine (AZA) or 6-mercaptopurine (6-MP) must be discontinued at least 2 weeks before inclusion into the study (Week 0 visit)
* Anti-TNF therapy in the 2 weeks before the Week 0 visit
* Failure of cyclosporine therapy in the previous 6 months prior to Screening visit
* Patients with serum albumin < 2.5 g/dl at baseline
* Low serum folate defined as decrease of >10% below normal range
* Patients with WBC< 3.0 x109th/L at baseline
* Patients with platelet count < 100 x109th/L
* Patients with an underlying infection with C. difficile at Screening visit
* Patients with pre-existing hepatic disease
* Patients with known non-alcoholic fatty liver disease (NAFLD)
* Patients with known Hepatitis B or Hepatitis C
* Patients with pre-existing renal dysfunction (creatinine >1.5 mg/dl).
* Patients with a pre-existing chronic lung disease other than well controlled asthma
* Patients with interstitial lung disease of unknown cause
* Patients with a BMI >35
* Known previous or concurrent malignancy (other than that considered surgically cured, with no evidence for recurrence for 5 years - basal cell does not exclude)
* Existing pregnancy, lactation, or planned pregnancy* (men and women) within the next 12 months. (*Methotrexate should not be used for at least 3 months before planned pregnancy for men and women and should not be used during pregnancy or breast feeding)
* High alcohol consumption (more than seven drinks per week)
* Non - steroidal inflammatory medications (NSAIDs) as long-term treatment, defined as use for at least 4 days a week each month
* Continuous treatment with one of the following drugs:
* Probenecid,
* Trimethoprim/sulfamethoxazole
* Sulfasalazine
* Acitretin
* Streptozocin
* Non-use of appropriate contraceptives in females of childbearing potential (e.g. condoms, intrauterine device {IUD}, hormonal contraception, or other means considered adequate by the responsible investigator) or in males with a child-fathering potential (condoms, or other means considered adequate by the responsible investigator during treatment
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial
* Well-founded doubt about the patient's cooperation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Herfarth, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (31):
- United States (31):
  - University of Southern California, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Shafran Gastroenterology, Winter Park, Florida
  - Atlanta Gastroenterology, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Indiana University IU Health, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Metropolitan Gastroenterology Group, PC, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Minnesota Gastroenterology, Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth College, Lebanon, New Hampshire
  - Mt Sinai School of Medicine, New York, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, Charlotte, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn State University, State College, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Herfarth HH, Osterman MT, Isaacs KL, Lewis JD, Sands BE. Efficacy of methotrexate in ulcerative colitis: failure or promise. Inflamm Bowel Dis. 2010 Aug;16(8):1421-30. doi: 10.1002/ibd.21246. PMID 20186931
- [Derived] Herfarth H, Barnes EL, Valentine JF, Hanson J, Higgins PDR, Isaacs KL, Jackson S, Osterman MT, Anton K, Ivanova A, Long MD, Martin C, Sandler RS, Abraham B, Cross RK, Dryden G, Fischer M, Harlan W, Levy C, McCabe R, Polyak S, Saha S, Williams E, Yajnik V, Serrano J, Sands BE, Lewis JD; Clinical Research Alliance of the Crohn's and Colitis Foundation. Methotrexate Is Not Superior to Placebo in Maintaining Steroid-Free Response or Remission in Ulcerative Colitis. Gastroenterology. 2018 Oct;155(4):1098-1108.e9. doi: 10.1053/j.gastro.2018.06.046. Epub 2018 Jun 30. PMID 29964043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 256 patients were assessed for eligibility between February 2012 and May 2016 at 37 sites across the US. 76 met exclusion criteria and one patient withdrew consent during screening.
Groups:
- Induction Period (Week 1-16): Steroid taper for 12 weeks and 25 mg MTX sq once weekly + 1 mg folic acid daily
- Methotrexate Maintenance (Week 17-48): 25 mg MTX sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine
- Placebo Maintenance (Week 17-48): Placebo sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine
Period: Induction Period (week1-16)
Arm/Group | Induction Period (Week 1-16) | Methotrexate Maintenance (Week 17-48) | Placebo Maintenance (Week 17-48)
Started | 179 | 0 | 0
Completed | 84 | 0 | 0
Not Completed | 95 | 0 | 0
Not completed — Lack of Efficacy | 70 | 0 | 0
Not completed — Adverse Event | 16 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Period: Maintenance Period Week
Arm/Group | Induction Period (Week 1-16) | Methotrexate Maintenance (Week 17-48) | Placebo Maintenance (Week 17-48)
Started (84 patients completed the induction period and were randomized to maintenance period) | 0 | 44 | 40
Completed | 0 | 15 | 16
Not Completed | 0 | 29 | 24
Not completed — Lack of Efficacy | 0 | 22 | 22
Not completed — Adverse Event | 0 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Induction Period (Week 1-16)
Number analyzed (Participants) | 179
Age, Continuous [Mean (Full Range); unit: years] | 42 [19 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 169
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 155
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 179
Calprotectin week 0 (Induction period) or week 16 (Maintenance period) [Mean (Standard Deviation); unit: mg/kg] | 612 (524)
Site of disease [Count of Participants; unit: Participants]
  Left colon | 86
  Pancolitis | 93

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival Week 17-48
Description: Relapse-free survival: Total week 48 Mayo score not exceeding 2 points, with all individual subscores not exceeding 1 point and relapse free survival defined by a numerical stable Mayo score throughout 32 weeks of maintenance therapy without increase of 3 or more points in the partial Mayo clinic score (excluding sigmoidoscopy) compared to the partial Mayo score of the individual patient at randomization at week 16 and no steroid use or other immunosuppressive medication throughout the 32 week maintenance period.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Methotrexate Maintenance (Week 17-48): 25 mg MTX sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine
  Methotrexate: Induction period (week 1-16) (Open label):
  25 mg MTX sq once weekly + Steroid taper + 1 mg folic acid daily
  Maintenance period (week 17-48) (Randomization):
  25 mg MTX sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine
- Placebo Maintenance (Week 17-48): Placebo sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine
  Methotrexate: Induction period (week 1-16) (Open label):
  25 mg MTX sq once weekly + Steroid taper + 1 mg folic acid daily
  Maintenance period (week 17-48) (Randomization):
  Placebo sq once weekly + 1 mg folic acid daily + 2.4 g mesalamine
Arm/Group | Methotrexate Maintenance (Week 17-48) | Placebo Maintenance (Week 17-48)
Number analyzed (Participants) | 44 | 40
Participants | 12 | 12

2. Secondary Outcome: Mucosal Healing at Week 48.
Description: Mucosal healing is defined as an absolute Mayo subscore for endoscopy of 0 or 1
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate Maintenance (Week 17-48) | Placebo Maintenance (Week 17-48)
Number analyzed (Participants) | 44 | 40
Participants | 12 | 12

3. Secondary Outcome: Relapse of Disease Between Week 17-48
Description: Relapse of disease in the Maintenance period as defined as an increase of 3 or more points in the partial Mayo clinic score (excluding sigmoidoscopy) with an absolute clinical Mayo score ≥ 4 or need for retreatment with steroids.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate Maintenance (Week 17-48) | Placebo Maintenance (Week 17-48)
Number analyzed (Participants) | 44 | 40
Participants | 29 | 25

4. Other Pre Specified Outcome: Calprotectin Levels <250 mcg/g Stool in Patients in Response or in Remission at Week 16 With Calprotectin Levels ≥ 250 mcg/g Stool at Screening
Description: Steroid free clinical remission as defined as a Mayo score of ≤ 2 points with no individual subscore exceeding 1 point or steroid free clinical response defined as a reduction from baseline in the clinical Mayo score of ≥ 2 points and at least 25%, with an accompanying decrease in the rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore of 0-1 point and a clinical Mayo score ≤5 and stool calprotectin levels <250 mcg/g stool at week 16 of the induction period in the subgroup of patients with calprotectin >250mcg/g stool at screening.
Time Frame: 16 weeks
Population: 134 /179 (75%) patients had a calprotectin value ≥ 250 mcg/g stool at screening.
Measure: Count of Participants; unit: Participants
Groups:
- Induction Period (Week 1-16): All patients treated with open label methotrexate 25 mg/kg bodyweight for 16 weeks in the Induction Period and a steroid taper week 0-12.
Arm/Group | Induction Period (Week 1-16)
Number analyzed (Participants) | 134
Participants | 56

5. Other Pre Specified Outcome: Calprotectin Levels <250 mcg/g Stool in Patients in Response or in Remission at Week 48 With Calprotectin Levels > 250 mcg/g Stool at Screening
Description: Steroid free clinical remission as defined as a Mayo score of ≤ 2 points with no individual subscore exceeding 1 point or steroid free clinical response defined as a reduction from baseline in the clinical Mayo score of ≥ 2 points and at least 25%, with an accompanying decrease in the rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore of 0-1 point and a clinical Mayo score ≤5 and stool calprotectin levels <250 mcg/g stool at week 32 of the maintenance period in the subgroup of patients with calprotectin ≥ 250mcg/g stool at screening.
Time Frame: 48 weeks
Population: 33/44 patient in the Methotrexate Maintenance group and 32/40 patients in the Placebo Maintenance group met the criteria of calprotectin ≥ 250 mcg/g stool at screening
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate Maintenance (Week 17-48) | Placebo Maintenance (Week 17-48)
Number analyzed (Participants) | 33 | 32
Participants | 10 | 8

6. Other Pre Specified Outcome: Calprotectin Levels < 50 mcg/g Stool in Patients in Remission at Week 16 With Calprotectin Levels ≥ 250 mcg/g Stool at Screening
Description: Steroid free clinical remission as a Mayo score of ≤ 2 points with no individual subscore exceeding 1 point and stool calprotectin levels of ≤ 50mcg at week 16 of the induction period in the subgroup of patients with calprotectin ≥ 250mcg/g stool at screening.
Time Frame: 16 weeks
Population: 134 /179 (75%) patients had a calprotectin value ≥ 250 mcg/g stool at screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period (Week 1-16)
Number analyzed (Participants) | 134
Participants | 10

7. Other Pre Specified Outcome: Calprotectin Levels < 50 mcg/g Stool in Patients in Remission at Week 48 With Calprotectin Levels ≥ 250 mcg/g Stool at Screening
Description: Steroid free clinical remission as a Mayo score of ≤ 2 points with no individual subscore exceeding 1 point and stool calprotectin levels of ≤ 50mcg at week 48 of the induction period in the subgroup of patients with calprotectin ≥ 250mcg/g stool at screening.
Time Frame: 48 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate Maintenance (Week 17-48) | Placebo Maintenance (Week 17-48)
Number analyzed (Participants) | 33 | 32
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: The adverse events were collected from each study participant from the screening visit until last study visit , which could be early termination or the last visit of the study (week 48).
Arm/Group | Induction Period (Week 1-16) | Methotrexate Maintenance (Week 17-48) | Placebo Maintenance (Week 17-48)
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/44 | 0/40
Serious Adverse Events (participants affected / at risk) | 15/179 | 0/44 | 1/40
Other Adverse Events (participants affected / at risk) | 69/179 | 41/44 | 30/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period (Week 1-16) (N=179) | Methotrexate Maintenance (Week 17-48) (N=44) | Placebo Maintenance (Week 17-48) (N=40)
Hospitalization (Gastrointestinal disorders) | 15 (18) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period (Week 1-16) (N=179) | Methotrexate Maintenance (Week 17-48) (N=44) | Placebo Maintenance (Week 17-48) (N=40)
Abdominal Discomfort (Gastrointestinal disorders) | 11 (13) | 13 (13) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 14 (14) | 13 (13)
Dizziness (Nervous system disorders) | 10 (11) | 1 (1) | 3 (3)
Elevated liver enzymes (Hepatobiliary disorders) | 6 (6) | 5 (5) | 3 (3)
Fatigue (Nervous system disorders) | 19 (20) | 5 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 36 (39) | 13 (16) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
There were no limitations for this trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT01393405/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT01393405/SAP_001.pdf